CLINICAL TRIAL: NCT04397159
Title: Objective and Subjective Measures of Fatigability in Veterans With Chronic Kidney Disease Before and After Flywheel Resistance Plus Aerobic Exercise
Brief Title: Effects of Combination Exercise on Fatigability in Veterans With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F3423-W
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Predialysis
Keywords: fatigability; strength; rehabilitation; eccentric exercise; combination exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Flywheel Resistance Plus Aerobic Exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Exercise (Experimental): Flywheel resistance exercise plus aerobic exercise
  Interventions: Behavioral: Combination Exercise
- Standard-of-care (No Intervention): Participants will maintain standard-of-care and current activity levels during the course of the study.

INTERVENTIONS:
Behavioral: Combination Exercise — Flywheel Resistance Plus Aerobic Exercise
  Other Names: Flywheel Resistance Plus Aerobic Exercise
  Arms: Combination Exercise

SUMMARY:
The VA health care system uses a health promotion-focused model which aims to provide longitudinal care through a patient-aligned care team for Veterans with chronic kidney disease. Since the largest subpopulation of Veterans with chronic kidney disease is comprised of those not requiring dialysis, neuromuscular screening assessments may provide valuable information regarding an individual overall health status and potential for future complications. Furthermore, identifying at risk individuals early in the disease process will allow for the prescription of timely interventions. Exercise strategies such as combination exercise, which uses flywheel resistance plus aerobic exercise, may provide a valuable treatment option for combating neuromuscular dysfunction and functional decline in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a complex medical condition affecting as much as 36% of the Veteran population. Both empirical and anecdotal evidence identify elevations in fatigability as a major health concern in Veterans with CKD predialysis. Neuromuscular deteriorations resulting from CKD are likely to contribute to excessive fatigability, impacting an individual's functional status. Flywheel resistance exercise (FRE) uses inertial resistance to allow for optimal muscle loading through the entire concentric muscle action and promotes greater eccentric force generation compared to traditional resistance exercise. FRE has been shown to be superior to traditional resistance exercise for improving muscle strength, power, and physical function in healthy populations suggesting it may be a useful treatment for addressing neuromuscular impairments and functional decline. However, it is unclear if the addition of aerobic exercise to FRE would provide additive improvements in fatigue resistance in patients with CKD, without compromising neuromuscular and functional benefits. The purpose of this project is to (1) advance the understanding of performance fatigability and perceived fatigability, and the association with neuromuscular capacity in Veterans with CKD stage 3 & 4 predialysis and (2) determine the extent to which combination FRE plus aerobic exercise training can improve fatigability status, neuromuscular capacity, and physical function in Veterans with CKD stage 3 & 4 predialysis. The central hypothesis is that reductions in neuromuscular capacity are associated with increases in fatigability severity, and that FRE plus aerobic exercise training will reduce fatigability severity while enhancing neuromuscular and functional capabilities in Veterans with CKD stage 3 & 4 predialysis. To address this hypothesis, researchers will characterize performance fatigability and perceived fatigability, and assess the associations between fatigability outcomes and neuromuscular capacity in Veterans with CKD stage 3 & 4 predialysis and examine the effects of 12-weeks of FRE plus aerobic exercise training on changes in performance and perceived fatigability, neuromuscular capacity, and physical function in Veterans with CKD stage 3 & 4 predialysis. Findings from this project will provide valuable information for advancing the understanding of performance fatigability and perceived fatigability, and their inter-relationship, in Veterans with CKD stages 3 and 4. Additionally, novel evidence on the responsiveness of performance and perceived fatigability, neuromuscular capacity, and quality of life to FRE plus aerobic exercise training will be gained.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory (with or without a gait aid), 50 years of age or older diagnosed with chronic kidney disease (CKD) stages 3 & 4 predialysis (as defined by eGFR 59-15 ml/min per 1.73m2)
* Control group will include ambulatory individuals without clinical evidence of kidney disease (defined by eGRF >60 ml/min per 1.73m2) within the last 12-months
* All participants must be able to speak and read English, and demonstrate orientation to person, place, and time

Exclusion Criteria:

* adults diagnosed with acute renal failure/injury within the last 12-months
* non-ambulatory individuals
* adults who do not use the DC VAMC as their main site for renal care
* those who have any uncontrolled cardiovascular
* musculoskeletal disease
* or other conditions that, in the opinion of the principal investigator, could make participation in the study unsafe
* any orthopedic or joint pain which would prevent the participant from safely engaging in the study protocol
* additionally, individuals with plans to relocate from the DC metro area within one year will not be eligible for the intervention portion of the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
change in knee extensor fatigability | week 6 and 12
  Knee extensor fatigability will be assessed as changes in torque of the dominant leg during 30 contractions.
change in perceived fatigability | week 6 and 12
  Rating of perceived fatigability will be assessed using a 10-point scale with 0 indicating "not fatigued at all" and 10 indicating "absolutely exhausted". Low scores reflect lower perceived fatigability.
change in muscle blood flow | week 6 and 12
  Muscle blood flow of the vastus lateralis will be assessed using near-infrared spectroscopy and determined as the change in total hemoglobin during venous occlusion test.

SECONDARY OUTCOMES:
change in muscle Quality | week 12
  Muscle quality of the vastus lateralis will be assessed using diagnostic ultrasound and determined using grayscale analysis.
change in Sit-to-Stand | week 12
  Sit-to-stand test will be used to assess physical function and determined as the time taken to complete five sit-to-stand repetitions.
change in rate of torque development | week 12
  Rate of torque development will be calculated as the change in torque over the change in time during isometric knee extensions.

OTHER OUTCOMES:
change in muscle activation | week 12
  Muscle activation of the vastus lateralis will be determined using electromyography as the root mean square during isometric knee extensions.
change in interleukin 6 (IL-6) and tumor necrosis factor alpha | week 12
  Interleukin 6 (IL-6) (pg/ml) and tumor necrosis factor alpha (pg/ml) will be assessed from blood samples.
change in health-related quality of life | week 12
  Health-related quality of life will be assessed using the Short-form 36
change in high density c-reactive protein | week 12
  Change in high density c-reactive protein (mg/L) will be assessed from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jared M. Gollie, PhD, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No